CLINICAL TRIAL: NCT02069327
Title: The Role of Fat Emboli in the Trauma Inflammatory Response
Status: Completed | Type: Observational
Sponsor: Poudre Valley Health System (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Principal Investigator, Julie Dunn, M.D., Trauma Research Director / Trauma Surgeon, Poudre Valley Health System
Other Study IDs: Fat Emboli
Record Dates: First submitted 2014-02-03; First posted 2014-02-24 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Femoral Fracture
Keywords: Femur; Fat; Emboli; Bone; Marrow; proteomic; proteomics; metabolomics; metabolomic; inflammatory; cytokine; chemokine; anaphlylatoxin; Thromboelastography; Medical Center of the Rockies; Fat Embolism Syndrome; Injury; Fracture; Metabolite; MCR; TEG; FES
MeSH Terms: conditions — Femoral Fractures; Platelet Glycoprotein IV Deficiency; Embolism; Embolism, Fat; Wounds and Injuries; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow Blood specimen (~4 teaspoons)
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study designed to investigate the role of fat emboli in patients who are undergoing a tibial or femoral fracture procedure in the operating room. The purpose of this study is to obtain samples of bone marrow and blood during tibial or femoral fracture procedures to understand the inflammatory response.

DETAILED DESCRIPTION:
Bone marrow is routinely removed during a tibial or femoral fracture procedure; researchers will take samples for this study from bone marrow that has already been removed as part of this procedure. No additional marrow samples will be taken as part of this research study. Also, researchers will collect blood (about 4 teaspoons) for testing inflammatory response and coagulation. Researchers may need to insert an additional line to collect your blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a tibial or femoral fracture procedure in the operating room.

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing a tibial or femoral fracture procedure in the operating room.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Inflammatory Response | One day
  Samples will be tested using proteomic and metabolomic assays from samples of bone marrow reamed during intramedullary (IM) femoral nailing.
  Blood samples drawn at the time of IM nailing will be tested to determine if clinically relevant amounts of marrow containing these inflammatory mediators are released into the bloodstream.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Dunn, M.D., Principal Investigator — Poudre Valley Health System
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States

IPD SHARING:
Plan to Share IPD: No